CLINICAL TRIAL: NCT05844267
Title: Sedentary Behavior With Physical Activity Breaks Aimed at Improving Cardiometabolic Risk Factors in Workers
Brief Title: Stand Up for Your Health: The Up Project
Acronym: TUP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Valparaiso (Other)
Responsible Party: Principal Investigator, Carlos Cristi Montero, Professor, School of Physical Education, Pontificia Universidad Católica de Valparaíso, Valparaíso, Chile, Pontificia Universidad Catolica de Valparaiso
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: BIOPUCV-HB 580-2023
Record Dates: First submitted 2023-04-24; First posted 2023-05-06 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Sedentary Behavior
Keywords: Sedentary time; Metabolic Health; Physical Activity; Body composition; Accelerometry
MeSH Terms: conditions — Sedentary Behavior; Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Booster Breaks group (led breaks) (Experimental): Participants will engage in active breaks led by a professional, where they will perform various exercises based on the guidelines provided by the Chilean safety association (ACHS). These breaks will have an average duration of 14-16 minutes per day and will take place from Monday to Friday for a period of 12 weeks.
  Interventions: Behavioral: Experimental led booster breaks
- Computer Prompts group (unled breaks) (Experimental): Active breaks will be guided by an application called "Ponte de Pie por tu Salud," designed by the Chilean Ministry of Health which will be installed on the participants' computers. The application will be configured to generate breaks every hour for a duration of 2 minutes for 8 hours, ensuring that an average of 14-16 minutes of active breaks are accumulated throughout the day.
  Interventions: Behavioral: Experimental unled computer-prompts
- Control (No Intervention): The group will participate in evaluations pre-post but not interventions. We will recommend continuing with their usual routine.

INTERVENTIONS:
Behavioral: Experimental led booster breaks — Participants in this group will receive interventions in the form of active breaks, administered by professionals in the relevant field, such as Physical Education teachers, for a period of 12 weeks. The active breaks will comprise exercises of light-to-moderate intensity, based on the guidelines provided by the Chilean safety association (ACHS), with an average duration of 14-16 minutes per day from Monday to Friday. The exercise types and progression will be elaborated in our protocol and published as supplementary material.
  Arms: Booster Breaks group (led breaks)
Behavioral: Experimental unled computer-prompts — Participants in this group will receive interventions in the form of active breaks, facilitated through an application called "Ponte de pie por tu salud," proposed by the Chilean Ministry of Health. This off-line application will be configured to generate breaks every hour, lasting for 2 minutes per break, over the course of 8 hours. This ensures that an average of 14-16 minutes of active breaks are accumulated throughout the day. Our research team will install the application on the participants' work computers and collect data from these computers weekly. At the end of the intervention period, the application will be uninstalled if necessary.
  Arms: Computer Prompts group (unled breaks)

SUMMARY:
In today's modern workplace, desk-based work is prevalent, leading to prolonged periods of sitting and limited physical activity among workers. This sedentary behavior can have detrimental effects on the physical and mental health of employees. Besides, this behavior contributes to the rising incidence of metabolic and general health problems in workers, even independently of their physical activity levels, leading to reduced productivity for the company and an increased economic burden on public health.

The Up Project is a Quasi-experimental controlled trial designed to assess the efficacy of two interventions to reduce sedentary behavior in the workplace. The study involves three groups: a) a control group, b) a group with booster breaks (led by professionals), and c) a group with unled computer prompts. The primary outcomes being measured are cardiometabolic risk and stress perception, while secondary outcomes include physical activity, sedentary behavior, and occupational pain.

This study is expected to contribute to the research gap in this area by providing valuable insights into the efficacy of interventions aimed at reducing sedentary behavior and its impact on health in the workplace.

DETAILED DESCRIPTION:
The design of The Up Project will be a Quasi-experimental controlled trial controlled trial in which participants will undergo two interventions aimed at reducing sedentary behavior in the workplace. The sample size was calculated using G*Power software and will consist of 60 workers from three higher education centers located in the Valparaiso region of Chile. Participants will be divided into three groups: a) a control group, b) a group with booster breaks led by professionals, and c) a group with computer prompts that are unled.

The study will be conducted in three stages, comprising two visits to our laboratory and one visit to the participants' offices. The first stage will involve a pre-intervention measurement session at our laboratory, which will comprehensively assess various cardiometabolic risk factors, such as body composition (DXA), waist circumference, weight, height, resting heart rate, and blood pressure. Questionnaires will also be administered to assess stress perception (PSS-14), occupational pain (using the Nordic-standardized questionnaire), physical activity (GPAQ), sedentary time at work (OSPAQ), 24-hour behavior (DABQ), eating habits (using the Mediterranean diet adherence questionnaire), smoking habits (using the Fargerstörm test), and socio-economic status (using the distribution and average autonomous income of households by income decile). Furthermore, participants will wear two types of accelerometers, ActiGraph and ActivPAL, for seven days to objectively measure physical activity intensity, sedentary time, and sedentary time breaks.

In the second stage, our research team will visit the participants' offices to remove the devices and administer the questionnaire application for sedentary time at work and 24-hour behavior for a second time. The intervention will commence after the accelerometers have been removed.

Finally, the third stage will involve a second visit to our laboratory, where cardiometabolic risk will be re-evaluated, and questionnaires on stress perception, occupational pain, physical activity, sedentary time at work, and 24-hour behavior will be administered again.

It is worth highlighting that mid-intervention, all three groups will be provided with accelerometers to re-evaluate the subjects' daily physical activity intensity, sedentary time, and breaks in sedentary time.

Intervention

The intervention will be conducted from Monday to Friday over a period of 12 weeks. The "Booster Breaks group" will receive a visit from a physical education teacher who will guide them through exercises based on the Chilean safety association (ACHS) guidelines. These exercises will last for an average of 14-16 minutes per day, and will be of light to moderate intensity, consistent with the intensity levels established during our pilot study.

The "Computer Prompts group" will have an offline messaging application ("Ponte de Pie por tu Salud") installed on their computers. The application will generate a message each hour, inviting the participants to stand up and perform exercises for 2 minutes. This will accumulate to an average of 14-16 minutes of active breaks daily. We will also be able to collect data on whether the participant rejected the break or proposed an alternative time.

It is important to note that both interventions will be equivalent in terms of intensity and time. The exercises for the "Booster Breaks group" will be performed at the same intensity and for the same duration (14-16 minutes) as the "Computer Prompts group." A detailed exercise plan for both groups can be found in the supplementary material.

The control group will only be evaluated pre and post-intervention and will be advised to continue with their usual routine.

Measurement of cardiometabolic risk factors:

Weight and Height: Weight was measured with a digital balance in which precision and maximum weight were of 0.1 and 150 kg respectively (OMROM. HN-289-LA). Height with a portable stadiometer (SECA, model 213, GmbH).

Body composition: Fat mass, fat-free mass, and bone mass will be assessed using a dual X-ray absorptiometer (General Electrics, model Lunar, series 212069). Both the equipment, box, and evaluators have been approved by the Health Service of the Region of Valparaiso.

Waist circumference: the minimum waist will be measured with a Lufkin metallic tape measure (W606PM) after exhaling.

Blood pressure: will be measured on the left arm with a digital monitor model HEM-7120 (OMRON, Illinois, USA) which provides both diastolic and systolic blood pressure values. It will be evaluated twice after 5 min of rest and the values will be averaged.

Resting heart rate: After the resting blood pressure assessment the minimum heart rate value will be recorded with a pulse oximeter model Prince-100B5 (Heal Force).

Measurement of physical activity and sedentary behavior:

Accelerometry: Time spent in sedentary and physical activity (and their intensities) will be objectively assessed with two accelerometers: the ActiGraph (Model GT3X+, Actigraph, Illinois, USA) and the ActivPAL ™ . Participants will use both devices for 7 consecutive days. The ActiGraph will be worn on the wrist, like a watch, which does not inconvenience one's routine tasks. It should only be removed for water activities (swimming) and showering. The ActivePAL is water-resistant and will be attached to the front of the right thigh with a hypoallergenic strap. Participants will also keep a monitoring diary to record how many times they used the accelerometers each day, the days they worked and the times they started and finished work on each of those days. Sleep quality will also be assessed with the GT3X+.

Self-reporting of physical activity: Global Physical Activity Questionnaire (GPAQ) is a questionnaire used by the World Health Organization to monitor physical activity levels worldwide (Bull et al., 2009).

Self-reporting of sedentary time at work: Occupational Sitting and Physical Activity Questionnaire (OSPAQ), allows the identification of the percentages of time the subject spends sitting down during the working day in which he/she works (Chau et al., 2012).

Self-reporting of behavior within 24 hours: Daily Activities Behavior Questionnaire (DABQ) allows the identification of the subject's behavior in terms of physical activity, sedentary time, and sleep in 24 hours (Kastelic et al., 2022).

Measurement of Stress Perceived Stress Scale Questionnaire (PSS-14): The questionnaire was originally developed and validated by Cohen, Kamarck, and Mermelstein in 1983. It has been adapted for use with Chilean adults and allows for the determination of an individual's stress level by scoring various domains related to stress tolerance using a Likert scale.

Measurement of Occupational Pain The Nordic standardized questionnaire will be used to assess the participants' perception of musculoskeletal symptoms related to their work. This questionnaire is a well-established tool for identifying and evaluating musculoskeletal problems and will allow us to gather information on any discomfort or pain experienced by the participants in their working environment. The questionnaire is designed to focus on the body areas most commonly affected by work-related musculoskeletal disorders, such as the neck, shoulders, back, and wrists. By using this questionnaire, we can identify any specific areas where participants may be experiencing pain or discomfort and tailor our intervention to address these issues (Kuorinka et al., 1987).

Measurement of Eating Habits Mediterranean diet adherence questionnaire. The questionnaire will be used to measure the subjects' adherence to the Mediterranean diet to determine its relationship with cardiometabolic factors (Martínez-González et al., 2012).

Measurement of smoking habits Fargerstörm test is a questionnaire that scores with a liker scale different aspects of smoking habits, which allows to determine the level of dependence to this substance (Heatherton et al., 1991).

Measurement of Socio-economic Status Distribution and average autonomous income of households by income decile. This questionnaire will be used to obtain the per capita income of the participants in order to have data on the socio-economic level of the subject. This questionnaire is made under the guidelines of the "Asesoria Tecnica Parlamentaria" of the Chilean government.

ELIGIBILITY:
Inclusion Criteria:

* Office workers who are physically and mentally healthy and work for 44 hours a week.

Exclusion Criteria:

* Individuals with physical limitations for physical exercise or undergoing weight loss treatment, pregnant women, or pacemaker users will be excluded.
* Participants who have another full-time job or part-time work in another job will also be excluded.
* Data from participants with a participation frequency of less than 70% in the physical activity sessions will not be considered.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-03-20 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Cardiometabolic Risk | up to six months
  Measurements related to cardiometabolic risk will be obtained through various methods, including DXA scans (General Electrics, model Lunar, series 212069) to determine body composition such as fat mass, fat-free mass, and bone mass. Weight will be measured in kilograms using a digital balance (OMRON HN-289-LA), height will be taken in centimeters with a portable stadiometer (SECA, model 213, GmbH). Additionally, weight and height will be combined to report BMI in kg/m^2. Waist circumference will be measured in centimeters using a Lufkin metallic tape measure (W606PM), while blood pressure will be measured in millimeters of mercury (mm Hg) using a digital monitor (model HEM-7120, OMRON) and heart rate will be measured in beats per minute using a pulse oximeter model Prince-100B5 (Heal Force).
Stress Perception | up to six months
  To measure stress perception, we will use the Perceived Stress Scale Questionnaire (PSS-14), which was validated by Cohen, Kamarck, and Mermelstein in 1983 and adapted for Chile by Erik Marín (Marín et al., 2004). The questionnaire assesses the individual's perception of various situations that may be influenced by their level of stress. The PSS-14 questions refer to the last month and are rated on a Likert scale ranging from 0 (never) to 4 (very often) in which a higher score indicates a higher level of perceived stress.

SECONDARY OUTCOMES:
Occupational pain | up to six months
  Measures of occupational pain will be obtained using the Nordic Musculoskeletal Questionnaire, a standardized tool recommended by the Institute of Public Health of the Chilean Ministry of Health. This questionnaire is designed to detect musculoskeletal symptoms related to desk-based work, including pain in the neck, shoulder, thoracic spine, wrist, lumbar spine, hip, knee, and ankle (Kuorinka et al., 1987). By using this tool, we will be able to assess both general and specific pain experienced by participants in the workplace. This questionnaire is answered with open and closed (yes/no) questions.
Physical Activity and Sedentary Time | up to six months
  Physical activity and sedentary time will be objectively measured in counts using two types of accelerometry: the ActiGraph (Model GT3X+, Actigraph, Illinois, USA) and the ActivPAL. Sleep quality will also be assessed using the ActiGraph GT3X+. Additionally, to measure physical activity in minutes, the Physical Activity Questionnaire (GPAQ) will be administered. This questionnaire is recognized by the World Health Organization (WHO) and is used to obtain information on the level of physical activity worldwide. To assess sedentary time, the Occupational Sitting and Physical Activity Questionnaire (OSPAQ) will be used to determine the sedentary time during work hours in percentage and frequency. Finally, the Daily Activities Behaviour Questionnaire (DABQ) will be administered to obtain information in minutes on subjects' physical activity, sedentary time, and sleep behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Cristi-Montero, Ph.D., Principal Investigator — Pontificia Universidad Católica de Valparaiso, Valparaiso,Chile
Locations (1):
- School of Physical Education, Pontificia Universidad Católica de Valparaíso, Valparaíso, Chile, Valparaíso, Región de Valparaíso, Chile